CLINICAL TRIAL: NCT07351656
Title: Screening for Heart Disease Using AI-Enabled Electrocardiography and Focused Cardiac Ultrasound: the AI CVD Screen Study.
Brief Title: A Study Of Heart Disease Using AI-Enabled Electrocardiography And Focused Cardiac Ultrasound
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul A. Friedman, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-012252
Record Dates: First submitted 2026-01-10; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Community dwelling adults (Experimental)
  Interventions: Diagnostic Test: Focused Cardiac Ultrasound; Diagnostic Test: 6-Lead AI-ECG; Diagnostic Test: 12-Lead AI-ECG
- Pregnant women (Experimental)
  Interventions: Diagnostic Test: Focused Cardiac Ultrasound; Diagnostic Test: 6-Lead AI-ECG; Diagnostic Test: 12-Lead AI-ECG
- Adolescents and young adults (Experimental)
  Interventions: Diagnostic Test: Focused Cardiac Ultrasound; Diagnostic Test: 6-Lead AI-ECG; Diagnostic Test: 12-Lead AI-ECG

INTERVENTIONS:
Diagnostic Test: Focused Cardiac Ultrasound — Focused cardiac ultrasound will utilize sonography to evaluate specific cardiac conditions, such as ventricular function, pericardial effusion, and valvular abnormalities.
Diagnostic Test: 6-Lead AI-ECG — A 6-lead ECG uses six electrodes placed on the chest and limbs to record the heart's electrical activity from multiple perspectives.
Diagnostic Test: 12-Lead AI-ECG — A standard 12-lead ECG consists of 12 leads: 6 limb leads and 6 chest (precordial) leads. These leads record the heart's electrical activity from different angles to provide a comprehensive assessment of cardiac function.

SUMMARY:
A study to evaluate feasibility, diagnostic yield, accuracy, and actionable thresholds of POC, immediate-feedback AI-ECG + AI FoCUS screening for cardiac disease in well described community populations.

ELIGIBILITY:
Adolescents and young adults:

Inclusion Criteria:

* Enrollment in a high-school, college or a resident in MN during the study period
* Age 15-29 years
* Informed consent (and assent for minors)

Exclusion Criteria:

* Presence of a pacemaker or defibrillator
* Inability to obtain a quality ECG tracing

Community dwelling adults:

Inclusion Criteria:

• Adult patients (>30 years of age, with pre-specified subgroups 30-64 and 65+))

Exclusion Criteria:

• Inability to provide informed consent to participate in the study

Pregnant women:

Inclusion Criteria:

* Adult female aged 18 to 49 years
* Pregnant at the time of enrollment
* Receiving obstetric care at identified study site(s)
* Willing and able to provide informed consent

Exclusion Criteria:

• Inability to provide consent

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19300 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with positive AI-ECG findings confirmed by echocardiography (Adolescents and young adults) | Baseline
  The percentage will be calculated as the number of participants whose AI-ECG results indicate a positive finding and are subsequently confirmed by echocardiography, divided by the total number of participants assessed, multiplied by 100.
Number of patients with positive AI-ECG detection for left-right sided SHD (Community Dwelling Adults) | Baseline
  Number of patients with positive AI-ECG detection for left-right sided SHD, defined as any of the following: LVEF <50%, >moderate right ventricular systolic dysfunction, >moderate aortic, mitral, or tricuspid valve regurgitation or stenosis, pulmonary hypertension (right ventricular systolic pressure > 50 mmHg), or elevated left-sided filling pressure.
Number of times the AI-ECG provides a correct diagnosis of clinically significant cardiac disease (Pregnant women) | Baseline
  Diagnostic performance of the AI-ECG will be determined by the accurate diagnosis of cardiomyopathy (left ventricular ejection fraction [LVEF] ≤50% or 10% or more decline in LVEF) or clinically significant structural heart disease (SHD; ≥ moderate right ventricular systolic dysfunction, ≥ moderate aortic, mitral, or tricuspid valve regurgitation or stenosis, pulmonary hypertension [right ventricular systolic pressure > 50 mmHg], or myocardial disease such as hypertrophic cardiomyopathy) in pregnant patients and those up to 6 weeks postpartum compared to standard of care.

SECONDARY OUTCOMES:
Number of false positive AI-ECG Results (Adolescents and young adults) | Baseline
  Number of false positive AI-ECG results will be determined by the number of positive AI-ECG results proven false from an echocardiography
Number of positive AI-ECG results for hypertrophic cardiomyopathy (HCM) (Adolescents and young adults) | Baseline
  The number of positive AI-ECG results for HCM will be based on how many patient ECGs indicate a possible diagnosis of HCM
Number of positive AI-ECG results for congenital heart defect (CHD) (Adolescents and young adults) | Baseline
  The number of positive AI-ECG results for CHD will be based on how many patient ECGs indicate a possible diagnosis of CHD
Proportion of patients by age group to receive a diagnosis (Community Dwelling Adults) | Baseline
  Proportion of patients by age group (30-39, 40-49, 50-65, 65-74, and 75 years and older) to receive a diagnosis from ultrasound that is confirmed by a comprehensive diagnostic work up.
Proportion of total patients to receive a diagnosis based on screening with 6 lead ECG (Community Dwelling Adults) | Baseline
  Proportion of total patients to receive a diagnosis based on screening with 6 lead ECG will be determined by the number of patients to have a correct diagnosis using the 6 lead ECG confirmed by echocardiogram compared to the total number of patients.
Proportion of total patients to receive a diagnosis based on screening with 12 lead ECG (Community Dwelling Adults) | Baseline
  Proportion of total patients to receive a diagnosis based on screening with 12 lead ECG will be determined by the number of patients to have a correct diagnosis using the 12 lead ECG confirmed by echocardiogram compared to the total number of patients.
Proportion of total patients to receive a diagnosis based on screening with 12 lead only AI-ECG with adjunctive FoCUS (Community Dwelling Adults) | Baseline
  Proportion of total patients to receive a diagnosis based on screening with 12 lead only AI-ECG with adjunctive FoCUS will be determined by the number of patients to have a correct diagnosis using the 12 lead ECG with adjunctive FoCUS confirmed by standard of care echocardiogram compared to the total number of patients.
Proportion of total patients to receive a diagnosis based on screening with 12 lead only AI-ECG without adjunctive FoCUS (Community Dwelling Adults) | Baseline
  Proportion of total patients to receive a diagnosis based on screening with 12 lead only AI-ECG without adjunctive FoCUS will be determined by the number of patients to have a correct diagnosis using the 12 lead ECG without adjunctive FoCUS confirmed by standard of care echocardiogram compared to the total number of patients.
Number of non-cardiac adverse events (Pregnant Women) | Baseline
  Number of non-cardiac adverse events can include hypertensive disorders of pregnancy (gestational hypertension, pre-eclampsia, eclampsia), preterm delivery, gestational diabetes, small for gestational age delivery, placental abruption, and pregnancy loss.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Friedman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No